CLINICAL TRIAL: NCT06957340
Title: Observation on the Therapeutic Effect of Low-Intensity Transcranial Ultrasound Stimulation Combined With Upper Limb Virtual Reality Training on Post-Stroke Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Mingyan Zhuang, Principal Investigator, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PJ2025-02-01
Record Dates: First submitted 2025-04-19; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Post Stroke Depression; Stroke
Keywords: stroke; post stroke depression; TUS
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sham TUS group (Sham Comparator): The sham group only underwent upper limb virtual reality training, with LITUS serving as a placebo.
  Interventions: Device: sham TUS
- TUS group (Experimental): Low-Intensity Transcranial Ultrasound Stimulation combined with Upper Limb Virtual Reality Training
  Interventions: Device: Low-Intensity Transcranial Ultrasound Stimulation

INTERVENTIONS:
Device: Low-Intensity Transcranial Ultrasound Stimulation — LITUS is conducted using the UE880C model from RuAo Medical Technology Co., Ltd. (Beijing). The parameters are set as follows:Frequency: 800(1+10%) kHz,Pulse repetition period: 25 ms,Duty cycle: 50%,Output power: 1.2 W,Maximum output power duration: 0.6 W,Effective sound intensity: 0.4 W/cm².During treatment, the patient is placed in a quiet room and asked to relax in a seated position. Three ultrasound probes are coated with a coupling agent and positioned on the patient's forehead.The total treatment duration is 20 minutes.
  The upper limb rehabilitation virtual training is used by the EM-BURT02-01 model from Eston.The affected limb is fixed to the robotic arm. Each treatment session consists of two virtual games (such as "Airplane Battle," "Mosquito Smasher," and other motion-based games).Each game lasts for 10 minutes, totaling 20 minutes of treatment. Treatment is administered 5 times a week.
  Arms: TUS group
Device: sham TUS — In the sham group, the machine only operates for 30 seconds, then stopping. Due to the physical characteristics of ultrasound, this stimulation cannot be perceived.Treatment is administered 5 times a week.
  Arms: sham TUS group

SUMMARY:
Abstract:

objective:To study whether post-stroke depression can be improved through low-intensity transcranial ultrasound stimulation combined with upper limb virtual reality training, explore its possible mechanisms, and provide new rehabilitation strategies for further treatment of post-stroke depression patients.

Methods:30 patients with PSD were selected as the subjects, and randomly divided into sham control group and combination treatment group according to computer randomization. Each group was 15 cases. The combined treatment group was subjected to LITUS, virtual reality upper limb training, routine medication and rehabilitation treatment. The control group only conducted virtual upper limb training, routine medication and rehabilitation treatment, and TUS was a false stimulation treatment.

Keywords:Ultrasoun,transcranial,ultrasound,stimulation,virtual reality,stroke,post-stroke depression

DETAILED DESCRIPTION:
Abbreviation：Transcranial Ultrasound Stimulation(TUS),low intensity focused ultrasound (LIFU),low intensity transcranial Ultrasound stimulation(LITUS),virtual reality(VR),post-stroke depression(PSD),Wolf Motor Function Test(WFMT),Patient Health Questionnaire-9(PSQ-9),Hamilton Depression Scale(HAMD),Pittsburgh sleep quality index(PSQI)

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were as follows:

  1. First-time stroke patients diagnosed with ischemic stroke via imaging techniques such as CT or MRI;
  2. Duration of the disease between 15 days and 6 months, with stable condition;Age between 18 and 75 years;
  3. Patients without severe intellectual, language comprehension, or behavioral impairments, capable of completing scale assessments, with an MMSE score of ≥24;
  4. Hemiplegia on one side and at least a 3rd-level seated balance, with Brunnstrom stage II or higher for the upper limb，able to perform movements with the assistance of the upper limb virtual reality training；
  5. No use of antidepressant medications in the past month, with PHQ-9 score≥10 and HAMA score≥17；
  6. Patients who are aware of the study details and have signed the informed consent form.

Exclusion Criteria:

* The exclusion criteria were as follows:

  1. Patients with metallic implants in the cranium or those with a pacemaker;
  2. Patients with unstable conditions, multiple brain infarctions, severe heart disease, or other significant organ conditions and complications, or a history of cancer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
WMFT | From enrollment to the end of treatment at 4 weeks
  Wolf Motor Function Score: The Wolf Motor Function Test (WMFT) is the internationally preferred scale widely used to assess the effectiveness of rehabilitation training in improving upper limb function. It consists of 15 assessment items, many of which involve upper limb movements commonly used in daily life, such as placing the forearm on a table, grip strength, and fine motor skills. Each item is scored on a 6-point scale ranging from 0 to 5 based on the patient's functional performance, with higher scores indicating better function. The total score is 75. This assessment method is simple, easy to administer, does not easily fatigue the patient, and is particularly suitable for evaluating hand and upper limb functional recovery in stroke patients.
PHQ-9 | From enrollment to the end of treatment at 4 weeks
  PHQ-9 (Patient Health Questionnaire-9): The PHQ-9 is a commonly used screening tool for depression. It is based on the nine diagnostic criteria from the DSM-V (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, developed by the American Psychiatric Association). The scale is used to assess whether an individual has depression and to determine the severity of the condition. It has good reliability and validity, and its assessment is simple, quick, and well-accepted by patients. The total score is 27, with higher scores indicating greater severity of depression.
HAMD | From enrollment to the end of treatment at 4 weeks
  The Hamilton Depression Rating Scale (HAMD) is one of the most widely used scales in clinical settings for assessing depressive states. Based on its assessment content, it has three versions; the HAMD-24 version is used here. This version includes multiple indicators such as mood, somatic symptoms, and sleep, allowing for an effective evaluation of the patient's functional improvement.

SECONDARY OUTCOMES:
PSQI | From enrollment to the end of treatment at 4 weeks
  Pittsburgh Sleep Quality Index (PSQI): The Pittsburgh Sleep Quality Index (PSQI) was developed in 1989 by Dr. Buysse and colleagues from the Department of Psychiatry at the University of Pittsburgh, USA. This scale is suitable for evaluating sleep quality in individuals with sleep and mental disorders, recording the patient's sleep quality over the past month. It consists of 19 items, which are scored and grouped into 7 components. Each component is rated from 0 to 3, with a total score of 21.
BDNF and 5-HT | From enrollment to the end of treatment at 4 weeks
  Blood samples were collected at 7 a.m. The blood was centrifuged at 3500 r/min for 10 minutes to separate the serum.ELISA was used to measure brain-derived neurotrophic factor (BDNF) and serotonin (5-HT) levels. The measurements were taken both before treatment and 28 days after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No